CLINICAL TRIAL: NCT04306705
Title: A Retrospective Study of Evaluating Safety and Efficacy of Tocilizumab Compared to Continuous Renal Replacement Therapy in Controlling CRS Triggered by COVID-19
Brief Title: Tocilizumab vs CRRT in Management of Cytokine Release Syndrome (CRS) in COVID-19
Acronym: TACOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Hubei Xinhua Hospital (Other); Wuhan No.1 Hospital (Other); Wuhan Central Hospital (Other)
Responsible Party: Principal Investigator, YIKAI YU, Clinical professor, Tongji Hospital
Other Study IDs: WHTJCOVID-19
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Covid-19; SARS; Cytokine Storm; Cytokine Release Syndrome; Tocilizumab
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — tocilizumab; Standard of Care; Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (3):
- Tocilizumab: Subjects received 8 mg/kg (body weight) Tocilizumab once in 100 ml 0.9% saline solution and administered intravenously within no less than 60 minutes. Tocilizumab was administered according to the local label.
  Interventions: Drug: Tocilizumab; Other: Standard of care
- Continuous Renal Replacement Therapy: Femoral vein catheterization was performed to complete continuous renal replacement therapy for consecutive 3 times or more.
  Interventions: Other: Standard of care; Procedure: Continuous renal replacement therapy
- Standard care: Standard of care therapy per local written policies or guidelines.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Tocilizumab — Administered as an intravenous infusion.
  Other Names: Actemra
  Groups: Tocilizumab
Other: Standard of care — Standard of care therapy per local written policies or guidelines and includes balancing of electrolytes and acid-base, the provision of enteral or parenteral nutrients support, antibiotics therapy, oxygen therapy and noninvasive ventilation.
Procedure: Continuous renal replacement therapy — Catheter insertion site is femoral vein.
  Groups: Continuous Renal Replacement Therapy

SUMMARY:
Some patients infected with the COVID-19 can develop uncontrolled immune response, leading to potentially life-threatening damage to lung tissue. Tocilizumab was first approved by the U.S. FDA in 2010 for rheumatoid arthritis and might now be used to treat serious COVID-19 patients with lung damage, according to China's National Health Commission updated its treatment guidelines in 7th version.Continuous Renal Replacement Therapy (CRRT) was recommended by China's National Health Commission treatment guidelines in 1st-7th version to control sever COVID-19 patients.

DETAILED DESCRIPTION:
Tocilizumab doesn't directly kill the novel coronavirus. It's known as an inhibitor of the receptor of interleukin 6 (IL-6), a pro-inflammatory cytokine. In the disease COVID-19, the body may respond to the pathogen by overproducing immune cells and their signaling molecules in a dangerous phenomenon called cytokine release storm.It has been recently speculated that IL-6 as a main culprit in that immune over activation among COVID-19 patients, hence the Tocilizumab clinical trial was initiated. In 2017, the FDA also approved Tocilizumab to treat cytokine release syndrome (CRS), a form of cytokine storm caused by CAR-T treatment. The investigator's hypothesis was that Tocilizumab would be associated with better clinical outcomes, such as decreased systemic inflammation, improved survival rate, better hemodynamic and improved of respiratory distress.Systemic inflammatory response syndrome was one of the main indications for treatment with CRRT. So it is clinically significant to compare the efficacy and safety of Tocilizumab and CRRT in management of CRS triggered by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Agrees to the collection of oropharyngeal or anal swabs and venous blood per protocol.
2. Male or non-pregnant female adult ≥18 years of age at time of enrollment.
3. Has laboratory-confirmed novel coronavirus infection as determined by polymerase chain reaction (PCR), or other commercial or public health assay in oropharyngeal or anal specimen within 72 hours prior to hospitalization.
4. Illness of any duration, and at least one of the following:

   1. Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   2. Clinical assessment (evidence of rales/crackles on physical examination) AND SpO2 ≤93% on room air, OR
   3. Requiring mechanical ventilation and/or supplemental oxygen, OR
   4. Sustained fever in the past 24 hours and unresponsive to NSAID or steroid
5. Serum IL-6 ≥3 times the upper limit of normal

Exclusion Criteria:

1. Alanine transaminase/aspartate transaminase (ALT/AST) > 5 times the upper limit of normal.
2. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. estimated glomerular filtration rate (eGFR) < 30 ml /min/1.73 m^2)
3. Hemoglobin<80 g/L
4. Leukocytes<2.0×10^9
5. Platelets<50×10^9
6. Pregnancy or breast feeding.
7. Anticipated transfer to another hospital which is not a study site within 72 hours.
8. Expected life span does not exceed 7 days.
9. Allergy to any study medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Laboratory (RT-PCR) confirmed infection with 2019-nCoV. Lung involvement confirmed with chest imaging Hospitalized with a SaO2/SPO2≤93% on room air or Pa02/Fi02 ratio <300mmHg and ≤14 days since illness onset.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Normalization of Fever and Oxygen Saturation Through Day 14 | First dose date up to 14 days
  This is a composite outcome measure. Criteria for fever normalization: Temperature < 36.6 °C armpit, < 37.2 °C oral sustained for at least 72 hours and criteria for oxygen normalization: peripheral capillary oxygen saturation (Sp02) > 94% sustained for at least 72 hours.

SECONDARY OUTCOMES:
Duration of hospitalization | Up to 28 days
  Measured in days
Proportion of Participants With Normalization of Fever Through Day 14 | First dose date up to 14 days
  Criteria for: Temperature < 36.6 °C armpit, < 37.2 °C oral, or < 37.8 °C rectal sustained for at least 72 hours.
Change from baseline in white blood cell and differential count | Day 1 through Day 28
  Blood routine test
Time to first negative in 2019 novel Corona virus RT-PCR test | Up to 28 days
  Oropharyngeal or anal swabs
All-cause mortality | up to 12 weeks
  Date and cause of death (if applicable).
Change from baseline in hsCRP | Day 1 through Day 28
  Serum hsCRP
Change from baseline in cytokines IL-1β, IL-10, sIL-2R, IL-6, IL-8 and TNF-α | Day 1 through Day 28
  Serum inflammatory cytokines
Change from baseline in proportion of CD4+CD3/CD8+CD3 T cells | Day 1 through Day 28 (if applicable)
  Flow cytometry for peripheral whole blood

CONTACTS AND LOCATIONS:
Overall Officials: SHAOXIAN HU, M.D, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China